CLINICAL TRIAL: NCT04349228
Title: Assessment of the Efficacy and Safety of Hydroxychloroquine (HCQ) Administered as a Prophylaxis for Health Professionals Exposed to COVID19 and Working in Medical Intensive Care Units, in Tunisia. Multicentric Randomized Comparative Study
Brief Title: Assessment of the Efficacy and Safety of (HCQ) as a Prophylaxis for COVID19 for Health Professionals
Acronym: COVID_2Pro
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: - Interest in the use of HCQ is controversial.
Sponsor: Abderrahmane Mami Hospital (Other)
Collaborators: Eshmoun Clinical Research Center (Network); Datametrix (Industry)
Responsible Party: Principal Investigator, Dr Jalila Ben Khelil, Head of department, Abderrahmane Mami Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ECC2020-03
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: COVID19; Sars-CoV2; Hydroxychloroquine; Prophylaxis; Healthcare Worker
Keywords: HCQ; prophylaxie; Healthcare Worker; Hydroxychloroquine; COVID19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Arm1:Hydroxychloroquine (HCQ) (200 mg / day) for at least 2 months or until potential contamination**.
  Arm2:Placebo (1 tablet/day) for at least 2 months or until potential contamination**.
  ** If the participant is contaminated (COVID19+), he or she will be followed up by telephone according to the study schedule.
Who Masked: Outcomes Assessor
Masking Description: As the trial is open-label and to preserve the validity of the trial, the measurement of the endpoint must be blinded by a third party (i.e., an evaluator who is not aware of the arm to which the patient has been assigned or the treatment the patient is receiving) using the PROBE ("Prospective Randomized Open Blinded Endpoint") method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine (HCQ) (Experimental): Exposed health care professionals working in the intensive care unit
  Interventions: Drug: Hydroxychloroquine (HCQ)
- Placebo (Placebo Comparator): Exposed health care professionals working in the intensive care unit
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine (HCQ) — Hydroxychloroquine (HCQ) 200mg/day
  Other Names: Plaquenil
  Arms: Hydroxychloroquine (HCQ)
Drug: Placebo oral tablet — Placebo of Hydroxychloroquine (HCQ) without any active substance
  Other Names: Placebo of Plaquenil
  Arms: Placebo

SUMMARY:
Assessment of the Efficacy and Safety of Hydroxychloroquine (HCQ) Administered as a Prophylaxis for Health Professionals Exposed to COVID19 and Working in Medical Intensive Care Units, in Tunisia. Multicentric, Randomized Comparative Study

DETAILED DESCRIPTION:
Interventional, Multicentric, Randomized Controlled Study in Two Parallel Groups of 530 Healthcare Professionals working in the Intensive Care Unit Exposed to Risk of COVID19 Infection Taking Hydroxychloroquine (HCQ) (200 mg/day) VS Placebo

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COVID-19 (-)
* Works in a medical intensive care unit exposed to COVID-19 infection
* 18 years old < age < 65 years old
* Having given written consent for their participation in the study.

Exclusion Criteria:

* Diagnosis of COVID-19+
* Retinopathies,
* Hydroxychloroquine or other prophylactic treatments for VIDOC19 within one month prior to inclusion and throughout the study.
* Hypersensitivity to chloroquine or hydroxychloroquine or 4-aminoquinolines or any of the other components of this drug,
* Contraindication to prophylactic use of chloroquine, e.g. liver failure, known epilepsy, creatinine clearance < 30 ml/min.
* Inability to be monitored during the trial period
* Pregnancy and breastfeeding
* Psoriasis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Symptomatic COVID(+) infection rate | 60 days
  * Clinical Examination: Symptomatic COVID(+) infection rate (from randomization to the onset of signs suggestive of Covid19 infection or to the end of the study at 60 days) The rate of COVID19 infections is defined by the occurrence of the clinical signs below:
  * Cough
  * Dyspnea
  * Fever
  * Myalgia
  * Arthralgia
  * Rhinorrhea
  * Anosmia
  * Asthenia, fatigability Confirmation of the above symptoms and COVID(+) PCR infection during the 60days treatment period.
  * Biological Examination :
  * Measurement of viral load
  * Ion, liver, kidney, haematological assessment
  * Electrical Examination: ECG

CONTACTS AND LOCATIONS:
Overall Officials: Jalila Ben Khelil, Pr, Principal Investigator — Hopital Abderrahmane Mami
Locations (1):
- Eshmoun Clinical Research Centre/ Hôpital Abderrahmane Mami-Ariana, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No